CLINICAL TRIAL: NCT02842866
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Adults Age 56 Years and Older
Brief Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Adults 56 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET49
Record Dates: First submitted 2016-07-15; First posted 2016-07-25 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; MenACYW conjugate vaccine; Menomune® - A/C/Y/W-135
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Healthy, adult participants aged greater than or equal to (≥) 56 years received a single dose of MenACYW Conjugate Vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 2: Menomune® Vaccine (Active Comparator): Healthy, adult participants aged ≥56 years received a single dose of Menomune®- A/C/Y/W-135 Vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide Vaccine, Groups A, C, Y, and W-135 Combined

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — 0.5 milliliter (mL), Intramuscular (IM), single dose on Day 0.
  Other Names: MenACYW conjugate vaccine
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal Polysaccharide Vaccine, Groups A, C, Y, and W-135 Combined — 0.5 mL, Subcutaneous (SC), single dose on Day 0.
  Other Names: Menomune® - A/C/Y/W-135
  Arms: Group 2: Menomune® Vaccine

SUMMARY:
The aim of the study was to demonstrate non-inferiority of immunogenicity and evaluate the safety of a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid conjugate vaccine (MenACYW conjugate vaccine) compared to a single dose of Meningococcal Polysaccharide Vaccine Serogroups A, C, Y, and W-135 Combined (Menomune® - A/C/Y/W-135) in adults 56 years of age and older in the United States.

Primary objective:

-To demonstrate the non-inferiority of the vaccine seroresponse to meningococcal serogroups A, C, Y, and W following the administration of a single dose of MenACYW conjugate vaccine compared to those observed following the administration of a single dose of Menomune® - A/C/Y/W-135.

Secondary objective:

-To compare the serum bactericidal assay using human complement (hSBA) antibody geometric mean titers of meningococcal serogroups A, C, Y, and W following the administration of MenACYW conjugate vaccine to those observed following the administration of Menomune® - A/C/Y/W-135.

Observational objectives:

* To describe antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA at baseline (before vaccination) and 30 days after vaccination with MenACYW conjugate vaccine or Menomune® - A/C/Y/W-135 in a subset of 100 participants per treatment group.
* To describe the safety profile of MenACYW conjugate vaccine compared to that of the licensed Menomune® - A/C/Y/W-135 after a single administration.

DETAILED DESCRIPTION:
Participants were randomized in a 1:1 ratio to receive a single dose of MenACYW conjugate vaccine or Menomune® - A/C/Y/W-135 on Day 0 (Visit 1).

Participants underwent immunogenicity assessment at baseline (pre-vaccination) and at 30 to 44 days post-vaccination and were also evaluated for safety up to Day 180 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥56 years on the day of inclusion.
* Informed consent form had been signed and dated.
* Attended all scheduled visits and complied with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (were considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination).
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceded the trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which might be received at least 2 weeks before or after study vaccine. This exception included monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B vaccine).
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to latex or any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within at least 10 years of the proposed study vaccination.
* Verbal report of thrombocytopenia, contraindicating IM vaccination, in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination in the Investigator's opinion.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >=100.4 degree [°] Fahrenheit [F]). A prospective participant was not included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (32):
- United States (31):
  - Chandler, Arizona
  - Anaheim, California
  - San Diego, California
  - Waterbury, Connecticut
  - Clearwater, Florida
  - DeLand, Florida
  - Jacksonville, Florida
  - Ponte Vedra, Florida
  - Port Orange, Florida
  - West Palm Beach, Florida
  - Lenexa, Kansas
  - Newton, Kansas
  - Wichita, Kansas
  - Elkridge, Maryland
  - Quincy, Massachusetts
  - Troy, Michigan
  - St Louis, Missouri
  - Endwell, New York
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Grants Pass, Oregon
  - Allentown, Pennsylvania
  - Uniontown, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Dallas, Texas
  - South Jordan, Utah
  - West Jordan, Utah
  - Charlottesville, Virginia
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Esteves-Jaramillo A, Koehler T, Jeanfreau R, Neveu D, Jordanov E, Singh Dhingra M. Immunogenicity and safety of a quadrivalent meningococcal tetanus toxoid-conjugate vaccine (MenACYW-TT) in >/=56-year-olds: A Phase III randomized study. Vaccine. 2020 Jun 9;38(28):4405-4411. doi: 10.1016/j.vaccine.2020.04.067. Epub 2020 May 6. PMID 32387012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from 15-July-2016 to 13-February-2017 at 35 sites in the United States and Puerto Rico.
Pre-assignment Details: Total 907 participants were enrolled in the study, out of which 906 were randomized. 1 participant was not randomized to either of the 2 treatment groups; this participant was not vaccinated and did not provide blood samples, therefore not counted in any analysis.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, adult participants aged greater than equal to (≥) 56 years received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid (MenACYW) Conjugate Vaccine on Day 0.
- Group 2: Menomune® Vaccine: Healthy, adult participants aged ≥56 years received a single dose of Meningococcal Polysaccharide Serogroups A, C, Y, and W-135 Combined (Menomune®) Vaccine on Day 0.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® Vaccine
Started (Randomized) | 451 | 455
Vaccinated | 448 | 453
Completed | 444 | 452
Not Completed | 7 | 3
Not completed — Serious Adverse Event | 0 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, adult participants aged ≥56 years received a single dose of MenACYW Conjugate vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® Vaccine | Total
Number analyzed (Participants) | 451 | 455 | 906
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (7.51) | 67.3 (7.53) | 67.1 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 261 | 520
  Male | 192 | 194 | 386
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 54 | 47 | 101
  White | 389 | 404 | 793
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Vaccine Seroresponse for Meningococcal Serogroups A, C, Y, and W Following Vaccination With Either MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: Vaccine seroresponse for serogroups A, C, Y, and W was measured by serum bactericidal assay using human complement (hSBA). It was defined as post-vaccination hSBA titers ≥1:16 for participants with pre-vaccination hSBA titers less than (<) 1:8, or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers ≥1:8.
Time Frame: Day 30 (Post-vaccination)
Population: Analysis was performed on per protocol analysis set which included all participants who received at least one dose of the study vaccine, had a valid post-vaccination serology result and had no protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® Vaccine
Number analyzed (Participants) | 433 | 431
percentage of participants
  Serogroup A | 58.2 [53.4 to 62.9] | 42.5 [37.7 to 47.3]
  Serogroup C | 77.1 [72.9 to 81.0] | 49.7 [44.8 to 54.5]
  Serogroup Y | 74.4 [70.0 to 78.4] | 43.4 [38.7 to 48.2]
  Serogroup W | 62.6 [57.8 to 67.2] | 44.8 [40.0 to 49.6]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup A; Test type: Non-Inferiority — The 95 percent (%) confidence internal (CI) of the difference in percentage was computed using the Wilson Score method without continuity correction. The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was greater than (>) -10 percent (%) for all four serogroups; Difference in percentage = 15.7, 95% CI 2-sided [9.08 to 22.2]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup C; Test type: Non-Inferiority — The 95% CI of the difference in percentage was computed using the Wilson Score method without continuity correction. The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for all four serogroups; Difference in percentage = 27.5, 95% CI 2-sided [21.2 to 33.5]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = 31.0, 95% CI 2-sided [24.6 to 37.0]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in percentage = 17.8, 95% CI 2-sided [11.2 to 24.2]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W were measured by hSBA method.
Time Frame: Day 30 (Post-vaccination)
Population: Analysis was performed on per-protocol analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilutions)
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® Vaccine
Number analyzed (Participants) | 433 | 431
titers (1/dilutions)
  Serogroup A | 55.1 [46.8 to 65.0] | 31.4 [26.9 to 36.7]
  Serogroup C | 101 [83.8 to 123] | 24.7 [20.7 to 29.5]
  Serogroup Y | 69.1 [58.7 to 81.4] | 21.0 [17.4 to 25.3]
  Serogroup W | 28.1 [23.7 to 33.3] | 15.5 [13.0 to 18.4]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup A; Test type: Other; GMT Ratio = 1.75, 95% CI 2-sided [1.40 to 2.20]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup C; Test type: Other; GMT Ratio = 4.10, 95% CI 2-sided [3.16 to 5.33]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup Y; Test type: Other; GMT Ratio = 3.30, 95% CI 2-sided [2.57 to 4.23]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Menomune® Vaccine; Serogroup W; Test type: Other; GMT Ratio = 1.81, 95% CI 2-sided [1.42 to 2.31]

ADVERSE EVENTS:
Time Frame: Unsolicited non-serious adverse events (AEs) were collected from Day 0 to Day 30 post-vaccination and solicited reactions (SR) were collected within 7 days post-vaccination. Serious Adverse Events were collected throughout the trial (up to 180 days post-vaccination).
Description: An SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was performed on safety analysis set which included participants who had received at least 1 dose of the study vaccine and have any safety data available.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® Vaccine
All-Cause Mortality (participants affected / at risk) | 0/448 | 2/453
Serious Adverse Events (participants affected / at risk) | 15/448 | 15/453
Other Adverse Events (participants affected / at risk) | 182/448 | 121/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=448) | Group 2: Menomune® Vaccine (N=453)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Column Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Device Failure (Product Issues) | 1 (1) | 0 (0)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=448) | Group 2: Menomune® Vaccine (N=453)
Injection Site Erythema (General disorders) | 23 (23) | 0 (0)
Injection Site Pain (General disorders) | 113 (113) | 43 (43)
Malaise (General disorders) | 65 (66) | 51 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 98 (100) | 69 (69)
Headache (Nervous system disorders) | 85 (85) | 66 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02842866/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT02842866/SAP_001.pdf